CLINICAL TRIAL: NCT02612766
Title: SAFETY AND TOLERABILITY OF OAT CONTAINING GLUTEN-FREE DIET
Acronym: SafeOatDiet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alfred Rusescu Institute for Mother and Child Care (Other)
Collaborators: The National Research and Development Institute for Alimentary Bioresources, Bucharest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCCA2-111/2012
Record Dates: First submitted 2015-11-11; First posted 2015-11-24 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Celiac Disease
Keywords: celiac disease; oat; gluten free diet
MeSH Terms: conditions — Celiac Disease; Gyrate Atrophy

ARMS (1):
- Single Arm (Other): This is a single-arm interventional study, in which each patient gets 50 grams/day of pure, uncontaminated oats
  Interventions: Dietary Supplement: Pure, uncontaminated oats

INTERVENTIONS:
Dietary Supplement: Pure, uncontaminated oats

SUMMARY:
The purpose of this study is to determine the safety and tolerability of oats in gluten free diet.

ELIGIBILITY:
Inclusion Criteria:

* Children over 4 years and adults with celiac disease (diagnosed according to current guidelines)
* Subject is able to fully participate in all aspects of this clinical trial

Exclusion Criteria:

* Known intolerance to oats
* Serious underlying disease other than CD which in the opinion of the investigator may interfere with the subject's ability to fully participate in the study

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in immunological activity of the disease measured by specific antibodies | After 6 weeks
Change in patient symptoms assessed by validated questionnaire | After 6 weeks

SECONDARY OUTCOMES:
Palatability of oat-containing gluten-free products is evaluated through a product liking questionnaire | After 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- "Alfred Rusescu" Institute for Mother and Child Care, Bucharest, Romania

REFERENCES:
- [Background] Kaukinen K, Collin P, Huhtala H, Maki M. Long-term consumption of oats in adult celiac disease patients. Nutrients. 2013 Nov 6;5(11):4380-9. doi: 10.3390/nu5114380. PMID 24201240
- [Background] Gatti S, Caporelli N, Galeazzi T, Francavilla R, Barbato M, Roggero P, Malamisura B, Iacono G, Budelli A, Gesuita R, Catassi C, Lionetti E. Oats in the diet of children with celiac disease: preliminary results of a double-blind, randomized, placebo-controlled multicenter Italian study. Nutrients. 2013 Nov 20;5(11):4653-64. doi: 10.3390/nu5114653. PMID 24264227
- [Background] Cooper SE, Kennedy NP, Mohamed BM, Abuzakouk M, Dunne J, Byrne G, McDonald G, Davies A, Edwards C, Kelly J, Feighery CF. Immunological indicators of coeliac disease activity are not altered by long-term oats challenge. Clin Exp Immunol. 2013 Mar;171(3):313-8. doi: 10.1111/cei.12014. PMID 23379438
- [Background] Tapsas D, Falth-Magnusson K, Hogberg L, Hammersjo JA, Hollen E. Swedish children with celiac disease comply well with a gluten-free diet, and most include oats without reporting any adverse effects: a long-term follow-up study. Nutr Res. 2014 May;34(5):436-41. doi: 10.1016/j.nutres.2014.04.006. Epub 2014 Apr 18. PMID 24916557
- [Background] Sjoberg V, Hollen E, Pietz G, Magnusson KE, Falth-Magnusson K, Sundstrom M, Holmgren Peterson K, Sandstrom O, Hernell O, Hammarstrom S, Hogberg L, Hammarstrom ML. Noncontaminated dietary oats may hamper normalization of the intestinal immune status in childhood celiac disease. Clin Transl Gastroenterol. 2014 Jun 26;5(6):e58. doi: 10.1038/ctg.2014.9. PMID 24964993
- [Background] Tjellstrom B, Stenhammar L, Sundqvist T, Falth-Magnusson K, Hollen E, Magnusson KE, Norin E, Midtvedt T, Hogberg L. The effects of oats on the function of gut microflora in children with coeliac disease. Aliment Pharmacol Ther. 2014 May;39(10):1156-60. doi: 10.1111/apt.12707. Epub 2014 Mar 24. PMID 24661128